CLINICAL TRIAL: NCT02318927
Title: A Responsive Closed-Loop Approach to Treat Freezing of Gait in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Medtronic (Industry); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB201400951
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Parkinsons Disease
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Deep Brain Stimulation (DBS) of Globus Pallidum plus Pedunculopontine Nucleus, including lead implant and battery placement. Magnetic Resonance Imaging and Computed Tomography (CT) scan will be obtained prior to implant. Measurement of number of Freezing of Gait (FoG) episodes during a FoG test at a lab. Other measures include freezing of gait questionnaire, gait and falls questionnaire, activities/balance confidence scale, Parkinson's disease quality of life questionnaire, Unified Parkinson's Disease Rating Scale physiology collection and sensor testing, adverse event recording, falls diaries, tracking use of assistive devices, gait and balance testing, and neuropsychological, neurosurgical, neurological, and physical exams.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation (DBS) of Globus Pallidum plus Pedunculopontine Nucleus, including lead implant and battery placement. Magnetic Resonance Imaging and Computed Tomography (CT) scan will be obtained prior to implant. Measurement of number of Freezing of Gait (FoG) episodes during a FoG test at a lab. Other measures include freezing of gait questionnaire, gait and falls questionnaire, activities/balance confidence scale, Parkinson's disease quality of life questionnaire, Unified Parkinson's Disease Rating Scale physiology collection and sensor testing, adverse event recording, falls diaries, tracking use of assistive devices, gait and balance testing, and neuropsychological, neurosurgical, neurological, and physical exams.

SUMMARY:
The study objective is to explore Deep Brain Stimulation (DBS) in two specific brain regions (Globus Pallidum, or GPI, plus the pedunculopontine nucleus, or PPN) for on medication freezing of gait (FoG) in Parkinsons Disease (PD). Hopefully, information gathered from these two brain regions after surgery will allow for the development of a personalized DBS system to address FoG. The primary outcome will be a comparison of the pre-operative number of FoG episodes in the laboratory during the FoG battery versus those 6 months post-DBS at the optimized device settings.

DETAILED DESCRIPTION:
As a participant in the study you will have the following procedure performed:

A series of questions by interview, questionnaires, and checklists will be collected. In addition, basic information (such as age, sex, race) and psychiatric, medical, and family history, physical and neurological exam that will include measuring vital signs (heart rate and blood pressure). There will be a "Falls Diary' to complete (an account of falling incidents and the details). Specific testing will be done to evaluate the gait and balance which will be repeated throughout the study. A psychiatric evaluation of mood and emotion will be performed including a detailed psychological testing, consisting of perception, learning, and memory. These psychological assessments will be repeated at every study visit. An MRI and a CT scan will be performed to make sure of the exact location of the DBS implant. The study will end in 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical diagnosis of idiopathic PD, without a previous DBS operation
2. Must be deemed appropriate for a GPi DBS operation by the interdisciplinary screening team (GPi must be the target chosen as most appropriate for treatment of their PD to qualify for this study)
3. Age 30-75 years (must meet UK Brain Bank criteria for diagnosis of idiopathic Parkinson's disease).
4. Experiencing significant gait and postural instability despite optimal pharmacologic management (Hoehn and Yahr Stage II or greater in the on state). 5. Best medication "on" does not reveal meaningful improvement in posture scores (Pull Test). Patients must be challenged in person with a suprathreshold dose of levodopa (1.5 times optimized regular dose of levodopa) and must have poor or no improvement in postural stability.

6. Patients must possess a clinical history of gait freezing > 2 episodes per month, to be included, participants must also score > 1 on item #3 of the Freezing of Gait (FOG) Questionnaire and exhibit five or more FoG episodes during the provocation protocol in on or off state.

7. L-dopa responsive with clearly defined "on" periods. 8. Willingness and ability to cooperate during conscious operative procedure, as well as during post-surgical evaluations, adjustments of medications and stimulator settings.

Exclusion Criteria:

1. Clinically significant medical disease that would increase the risk of developing pre- or postoperative complications. Clinically significant medical disease includes uncontrolled systemic hypertension with values above 170/100mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation which cannot be interrupted; any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.
2. Evidence of secondary or atypical parkinsonism.
3. Other neurological and musculoskeletal impairments that would negatively influence postural stability
4. Past MRI scan with significant evidence of brain atrophy or other abnormalities. 5. Dementia as evidenced by impairment in two neuropsychological domains and a Mattis Dementia Score <130.

6. A major untreated psychiatric disorder as revealed on psychiatric exam at screening, and a Beck Depression Inventory Score >14.

7. Subjects with a history of seizures. 8. Subjects who may require repeat MRI scans. 9. Subjects with a history of a cranial neurosurgical procedure. 10. Subjects with metal in the head or another implanted stimulator (e.g. vagus nerve stimulator, spinal cord stimulator, pacemaker, cochlear implant, etc).

11. Subjects who require treatment with Electroconvulsive therapy (ECT) or repetitive Transcranial Magnetic Stimulation (rTMS).

12. Pregnant or nursing women or women who wish to become pregnant will be excluded.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-11-03 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Number of Freezing of Gait (FoG) episodes in the laboratory during the FoG battery | Change from Baseline to 6 Months

SECONDARY OUTCOMES:
Number of adverse events (AE's) . | Change from Baseline to 24 Months
  The DSMB will review all adverse events (AE's) in real time. The device related AE definition will include both therapy and procedure related AE's. The Data Safety Monitoring Board (DSMB) will evaluate the study at least every 6 months and have the power to terminate the study for safety reasons.

OTHER OUTCOMES:
Freezing of gait questionnaire | Change from Baseline to 6 Months
Gait and falls questionnaire | Change from Baseline to 6 Months
Activities/balance confidence scale | Change from Baseline to 6 Months
Parkinson's disease quality of life questionnaire | Change from Baseline to 6 Months
Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 to assess Parkinson's disease symptom severity on medication and on stimulation | Change from Screening to 6 Months
Number of falls reported on Falls Diary | Change from Baseline to 6 Months
Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 to assess Parkinson's disease symptom severity off medication and on stimulation | Change from Screening to 6 Months
Total Unified Parkinson's Disease Rating Scale (UPDRS) to assess Parkinson's disease symptom severity on medication and on stimulation | Change from Screening to 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Okun, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States

REFERENCES:
- [Derived] Molina R, Hass CJ, Sowalsky K, Schmitt AC, Opri E, Roper JA, Martinez-Ramirez D, Hess CW, Foote KD, Okun MS, Gunduz A. Neurophysiological Correlates of Gait in the Human Basal Ganglia and the PPN Region in Parkinson's Disease. Front Hum Neurosci. 2020 Jun 4;14:194. doi: 10.3389/fnhum.2020.00194. eCollection 2020. PMID 32581744
- [Derived] Tahafchi P, Molina R, Roper JA, Sowalsky K, Hass CJ, Gunduz A, Okun MS, Judy JW. Freezing-of-Gait detection using temporal, spatial, and physiological features with a support-vector-machine classifier. Annu Int Conf IEEE Eng Med Biol Soc. 2017 Jul;2017:2867-2870. doi: 10.1109/EMBC.2017.8037455. PMID 29060496